CLINICAL TRIAL: NCT02798666
Title: High-intensity Interval Training is Associated With Greater Impact on Physical Fitness, Insulin Sensitivity and Muscle Mitochondrial Content in Overweight Males, as Opposed to Continuous Endurance Training: a Randomized Controlled Trial.
Brief Title: Effect of High-intensity Interval Training on Metabolic Fitness in Overweight Males.
Acronym: CALIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CALIN-001
Record Dates: First submitted 2016-05-31; First posted 2016-06-14 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Overweight and Obesity
Keywords: Physical fitness; Respiratory exchange ratio; Insulin sensitivity; High intensity interval training; Continuous exercise training
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity exercise training (Experimental): The participants exercised for 40 minutes, twice a week, under supervision of two physiotherapists for in total 10 weeks. Each training session included a warming up, a sprint interval block [10 minutes], continuous aerobic exercise [10 minutes], another sprint interval block [10 minutes] and cooling down. For the first 5 weeks, each sprint interval block consisted of 10 sprint bouts [>100 r/min] of 15 seconds at a cycling resistance matching with the ventilatory threshold [VTR], alternated with 45 seconds relative rest [50 r/min at VTR]. Starting from week 6 until week 10, the intensity of sprinting and relative rest was increased up to 110% of VTR.
  Interventions: Other: High intensity exercise training
- Continuous exercise training (Active Comparator): The comparative group performed a continuous aerobic training [CAT] for 10 weeks, twice a week and 40 minutes per session [volume and frequency is equal to HIIT]. The protocol of the CAT group consisted of warming up [stretching of the large muscle groups and cardiovascular exercises at 30% of peak cycling power output for five minutes], continuous aerobic exercise training [3 times 10 minutes] and cooling down [stretching of the large muscle groups and cardiovascular exercises at 30% of peak cycling power output for five minutes]. During the continuous aerobic protocol [cycling or stepping] participants exercised for 10 minutes at a HR similar to the HR at VT [60 r/min], which was increased to 110% of VT from week 6 onwards.
  Interventions: Other: Continuous exercise training

INTERVENTIONS:
Other: High intensity exercise training — Exercise training using sprint interval exercise
  Other Names: HIT
  Arms: High intensity exercise training
Other: Continuous exercise training — Exercise training using continuous exercise at constant heart rate
  Other Names: CAT
  Arms: Continuous exercise training

SUMMARY:
Background and aims: The purpose of this study was to evaluate the effect of high intensity interval training (HIIT) on body composition, physical fitness, metabolic fitness and muscle histology in men with overweight or obesity compared to continuous aerobic training (CAT).

Material and methods: 16 male participants with overweight/obesity (age range: 42 - 57 years, body mass index: 28 - 36 kg/m²) were randomized to HITT (n=8) or CAT (n=8). HIIT was composed of two sprint blocks of 10 minutes at ventilatory threshold (VT), within between a continuous block of 10 minutes, twice a week for 15 weeks. CAT was composed of three blocks of 10 minutes continuous endurance training at VT. After 5 weeks, intensity was increased to 110% of VT. Changes in body composition, physical fitness (peakVO2 and anaerobic threshold (AT)), basal respiratory exchange ratio (bRER) and insulin sensitivity by oral glucose tolerance test were evaluated. Mitochondrial content was evaluated by transmission electron microscopy (TEM) in muscle biopsies.

DETAILED DESCRIPTION:
Participants:

For this study, 16 adult males with overweight or obesity (BMI-range 28 - 36 kg/m2) were recruited and randomized in two experimental groups (high intensity training (n=8) and continuous moderate-intense aerobic training (n=8)). Randomization was done with the envelope method. Participants were excluded if they had diabetes (HbA1c>6,5%), severe musculoskeletal (eg osteoarthritis), cardiovascular (eg chronic heart failure) or respiratory (eg chronic obstructive pulmonary disease (COPD)) problems, based on medical files A signed informed consent was provided by all participants before study admission. The study was approved by the ethics committee of the Ghent University Hospital (B670201318620).

Intervention:

The intervention group performed a high intensity interval training [HIIT]. The HIIT group followed a 10-week training program. The participants exercised for 40 minutes, twice a week, under supervision of two physiotherapists. Each training session included a warming up [stretching of the large muscle groups and cardiovascular exercises at 30% of peak cycling power output for five minutes], a sprint interval block [10 minutes], continuous aerobic exercise [10 minutes], another sprint interval block [10 minutes] and cooling down [stretching of the large muscle groups and cardiovascular exercises at 30% of peak Watt for 5 minutes]. For the first 5 weeks, each sprint interval block consisted of 10 sprint bouts [>100 r/min] of 15 seconds at a cycling resistance matching with the ventilatory threshold [VTR], alternated with 45 seconds relative rest [50 r/min at VTR]. Starting from week 6 until week 10, the intensity of sprinting and relative rest was increased up to 110% of VTR.

Comparative group:

The comparative group performed a continuous aerobic training [CAT] for 10 weeks, twice a week and 40 minutes per session [volume and frequency is equal to HIIT]. The protocol of the CAT group consisted of warming up [stretching of the large muscle groups and cardiovascular exercises at 30% of peak cycling power output for five minutes], continuous aerobic exercise training [3 times 10 minutes] and cooling down [stretching of the large muscle groups and cardiovascular exercises at 30% of peak cycling power output for five minutes]. During the continuous aerobic protocol [cycling or stepping] participants exercised for 10 minutes at a HR similar to the HR at VT [60 r/min], which was increased to 110% of VT from week 6 onwards. The training was supervised by two physiotherapists.

In both exercise modes the participants cycled in the first and third block and cycled or stepped in the second block. The training programs were conducted in the Physiotherapy Department of the University Hospital of Ghent.

Outcome variables:

The quantification of all examined variables was performed by blinded assessors. All tests and measurements were conducted at the exercise laboratory of the Physiotherapy Department, Ghent University (maximal exercise test, metabolic flexibility) or at the Department of Endocrinology University Hospital Ghent (OGTT and muscle biopsy) or Department of Pathological Anatomy (muscle histology). Prior to all tests and measurements, participants were well informed and familiarized with the equipment and testing protocols. All participants from each group were tested on the same moment of day pre- and post-intervention. All participants maintained normal physical activity and dietary patterns, and refrained from exhaustive physical exercise three days prior to each experimental day Anthropometry Height was measured to the nearest 0.1 cm using a stadiometer (Holtain Ltd, Pembrokeshire, UK). Weight was measured to the nearest 0.1 kg on a digital balance scale (Seca, Germany) with the subject wearing lightweight clothing and no shoes. The body mass index (BMI) was calculated from weight and height.

Physical fitness Maximal cardiopulmonary exercise test. Participants were tested on a computer-driven cyclo-ergometer (Marquette Case, Marquette Electronics, Milwaukee, WI, USA) using a ramped protocol (20 W/ min) starting at 40 W. Twelve-lead electrocardiogram and heart rate (HR ) were recorded continuously during the test, whereas blood pressure was measured with a manual sphygmomanometer every two minutes. Subjects were familiarized with the test procedure before baseline testing. Subjects were asked and encouraged to perform exercise testing until physical exhaustion or until the physician stopped the test because of severe adverse events, such as increasing chest pain, dizziness, potentially life threatening arrhythmias, clinically important ST-segment deviations, marked systolic hypotension or hypertension. Tests were classified as maximal when respiratory exchange ratio (RER) increased above1.1. Respiratory gas measurements were obtained by using a Metalyzer 3B (Cortex, Leipzig, Germany). Oxygen consumption (VO2), carbon dioxide production (VCO2), minute ventilation (VE), tidal volume, respiratory rate and mixed expiratory carbon dioxide concentration were measured continuously with mixed chamber analysis. Peak VO2 was expressed as the highest attained VO2 during the final 30 seconds of exercise according to the American Thoracic Society guidelines. The ventilator threshold (VT) was determined based on the metabolic equivalents of O2 and CO2 (VE/VO2 and VE/VCO2). The point at which the VE/VO2 increased without an increase in VE/VCO2 was identified as the VT.

Basal respiratory exchange ratio Participants had to lie supine for 30 minutes after an overnight fast in a quiet and thermo-neutral environment. Basal oxygen consumption and carbon dioxide production was measured with an automated respiratory gas analyzer using a mask (Metalyzer 3B; Cortex, Leipzig, Germany). The gas analyzer system was calibrated before every experiment. RER was calculated as VCO2/VO2. This ratio lies in an interval between 0,7 en 1,0 indicating dominant fat oxidation to dominant carbohydrate oxidation.

Oral glucose tolerance test (OGTT) At 8:00 A.M. , after a 10- to 12-h overnight fast, subjects received a 75-g OGTT. Blood samples were taken at -30, -15, 0, 30, 60, 90, and 120 min for the measurement of plasma glucose and insulin concentrations. Insulin levels were determined using the immunoanalyzer COBAS e411 (Roche). Glucose was analysed by the hexokinase method (COBAS, Roche).

To evaluate insulin sensitivity an OGTT-composite score was calculation based on the reference of Matsudoa et al.. This score is composed as 10,000/square root of (fasting glucose x fasting insulin) x (mean glucose x mean insulin during OGTT). The higher the score, the better the insulin sensitivity.

Muscle biopsy After a 1-h rest period, a percutaneous needle biopsy sample was taken from the right vastus lateralis muscle with a biopsy gun (needle 14G) under local anesthetic through a 2-mm incision in the skin (2-3 ml lidocaine) under the guidance of echography. Two muscle samples of 15 mg were taken and incubated in PG (Paraformaldehyde and Glutaaraldehyde) for transmission electron microscopy (TEM).

Transmission Electron Microscopy TEM was used to determine IMCL and mitochondrial characteristics. Samples were viewed at 6,500× using a JEOL 1200EX TEM. Sixteen micrographs were acquired from 8 randomly sampled longitudinal sections of muscle fibers (2 micrographs/fiber) from each individual muscle - one micrograph acquired near the cell surface representing the subsarcolemmal (SS) region and the other acquired of parallel bundles of myofibrils representing the intramyofibrillar (IMF) region. Lipid droplets and mitochondrial fragments were circled and converted to actual size using a calibration grid. For each set of 16 images, mean IMCL or mitochondrial size (µm2), total number of IMCL droplets or mitochondria per square micrometer of tissue (#/µm2) were calculated in the IMF and SS compartments by digital imaging software (Image Pro Plus, ver. 4.0; Media Cybernetics, Silver Springs, MD). The reference for SS space quantification was the cytoplasmic space between the sarcolemma and the first layer of myofibrils.

Statistical analyses All data were analysed with a commercially available statistical software program (Statistical Package for the Social Sciences, SPSS 20.0, SPSS Chicago, IL, USA). Data are expressed as mean and standard deviation (SD). Due to the small sample size a non-parametric statistical evaluation was preferred. To evaluate pre-post differences within groups, a Wilcoxon test was performed. To evaluate pre-post differences between groups, differences between pre- and post-evaluation were calculated (pre minus post) and compared with a Mann Withney U test. Significance levels were set at P<0,05 for both tests. For the between group differences effect sizes were calculated based on Cohen's d values.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27 and 35

Exclusion Criteria:

* Diabetes (HbA1c>6,5%),
* severe musculoskeletal (eg osteoarthritis),
* cardiovascular (eg chronic heart failure) or respiratory (eg chronic obstructive pulmonary disease (COPD)) problems based on medical files.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity measured by oral glucose tolerance test | Baseline and 10 weeks (end of intervention)

SECONDARY OUTCOMES:
Respiratory exchange ratio measured by ergospirometry at rest | Baseline and 10 weeks (end of intervention)
muscle fiber fat content measured by transmission electron microscopy in muscle biopsy | Baseline and 10 weeks (end of intervention)
muscle fiber mitochondrial content measured by transmission electron microscopy in muscle biopsy | Baseline and 10 weeks (end of intervention)
PeakVO2 measured by ergospirometry during maximal exercise testing | Baseline and 10 weeks (end of intervention)
Ventilatory threshold measured by ergospirometry during maximal exercise testing | Baseline and 10 weeks (end of intervention)

OTHER OUTCOMES:
Weight measured by weight scale | Baseline and 10 weeks (end of intervention)
Heigth measured by stadiometer | Baseline and 10 weeks (end of intervention)
BMI | Baseline and 10 weeks (end of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Calders, Professor, Principal Investigator — Department of Rehabilitation Sciences and Physiotherapy, Universtity of Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cochran AJ, Percival ME, Tricarico S, Little JP, Cermak N, Gillen JB, Tarnopolsky MA, Gibala MJ. Intermittent and continuous high-intensity exercise training induce similar acute but different chronic muscle adaptations. Exp Physiol. 2014 May 1;99(5):782-91. doi: 10.1113/expphysiol.2013.077453. Epub 2014 Feb 14. PMID 24532598